CLINICAL TRIAL: NCT06570538
Title: Analgesic Efficacy of an Opioid-free Postoperative Pain Management Strategy Versus a Conventional Opioid-based Strategy Following Video-assisted Thoracoscopic Lobectomy: an Open-label, Randomized, Controlled, Non-inferiority Trial
Brief Title: Analgesic Efficacy of an Opioid-free Postoperative Pain Management Strategy Versus a Conventional Opioid-based Strategy Following Video-assisted Thoracoscopic Lobectomy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATHGuangzhou.
Record Dates: First submitted 2024-07-29; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain
Keywords: Lung Cancer; Postoperative pain; OFA; Erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Masking Description: In view of ethical considerations, the study was not blinded to anesthesiologists and patients, and the investigator responsible for postoperative follow-up was not involved in intraoperative anesthesia management.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB Group (Experimental): The drug composition of the analgesic pump for erector spinae block was 300 mL of 0.25% ropivacaine, the mode was intermittent pumping, and the parameters were set as follows: 30 mL of the first dose, 5 mL/h of the background dose, and 10 mL of the pumping every 6h for the first 24 hours after the operation.
  Interventions: Drug: Ropivacaine
- Convention group (Active Comparator): Intravenous analgesic is sufentanil ( 2.0 μg/kg), 0.9% saline diluted to 100 mL, background dose of 2 ml/h, no loading dose, activated after extubation and continued until 48 hours postoperatively.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Ropivacaine — 300 mL of 0.25% ropivacaine, the mode was intermittent pumping, and the parameters were set as follows: 30 mL of the first dose, 5 mL/h of the background dose, and 10 mL of the pumping every 6h for the first 24 hours after the operation.
  Other Names: Erector spinae plane block
  Arms: ESPB Group
Drug: Sufentanil — Sufentanil 2.0 μg/kg, 0.9% saline diluted to 100 mL, background dose of 2 ml/h, no loading dose, activated after extubation and continued until 48 hours postoperatively.
  Other Names: Intravenous analgesia
  Arms: Convention group

SUMMARY:
Investigators have designed a randomized controlled trial. Utilizing an open-label, randomized, controlled study methodology, this trial aims to explore a opioid-free, safe, and effective analgesic approach for thoracic surgery. It also seeks to provide clinical guidance for the implementation of opioid-free or reduced-opioid postoperative analgesia in other thoracic procedures, aiming to optimize postoperative pain management for patients and ultimately enhance the overall patients recovery experience.

DETAILED DESCRIPTION:
Patients who undergo thoracoscopic lobectomy are often at an elevated risk of opioid-related complications due to their reliance on opioids. This overdependence not only decelerates the postoperative recovery process but also significantly increases healthcare costs. Although there is a surge of interest in opioid-free anesthetic analgesia (OFA) for its potential to reduce adverse outcomes associated with opioid use, there is a dearth of randomized controlled trials examining the efficacy of postoperative analgesia in patients undergoing thoracoscopic surgery. Consequently, the actual effectiveness of OFA in improving postoperative pulmonary complications and facilitating patient recovery remains unclear. Its application is still in the exploratory phase, with clinical practice lacking definitive guidelines to endorse or discard OFA as an alternative for postoperative analgesia in thoracoscopic surgery.

To bridge this knowledge gap and evaluate the perioperative analgesic efficacy of OFA compared to traditionally used opioids in selected cancer patients undergoing thoracoscopic surgery, investigators have designed a randomized controlled trial. Utilizing an open-label, randomized, controlled study methodology, this trial aims to explore a opioid-free, safe, and effective analgesic approach for thoracic surgery. It also seeks to provide clinical guidance for the implementation of opioid-free or reduced-opioid postoperative analgesia in other thoracic procedures, aiming to optimize postoperative pain management for patients and ultimately enhance the overall patient recovery experience.

ELIGIBILITY:
Inclusion criteria:

* Aged between 18 and 65 years.
* Patients with lung cancer or suspected lung cancer who are undergoing lobectomy surgery via Video-assisted thoracoscopic surgery (VATS) or Robotic-assisted thoracoscopic surgery (RATS).
* American anesthesiologist association (ASA) physical status classificationⅠ-Ⅲ.
* Surgery is expected to last at least 2 hours, with a minimum of 2 days of postoperative hospitalization.
* Patients participate voluntarily and have signed an informed consent form.

Exclusion Criteria:

* Patients who underwent open-heart surgery.
* Patients with BMI ≥30 kg/m², or ≤18.5 kg/m².
* Patients who are allergic to any of the local anesthetic drugs, such as ropivacaine, lidocaine, bupivacaine, procaine, bupivacaine, benzocaine, dacronin, etc.
* Patients who are allergic to any of the general anesthesia drugs, such as those including propofol, sufentanil, remifentanil, etc.
* Patients who currently have active ulcers or have gastrointestinal bleeding or who are allergic to any NSAIDs such as parecoxib sodium, flurbiprofenol ester, and acetaminophen.
* Patients with contraindications to epidural spinal plane block (ESPB), such as skin infection near the puncture site or coagulation disorders.
* Patients allergic to ultrasound gel.
* Patients with significant preoperative renal insufficiency (creatinine more than twice the upper limit of normal).
* Patients with severe spinal deformities prior to surgery.
* Patients with preoperative distant tumor metastasis.
* Patients who have experienced cardiovascular or cerebrovascular accidents within the past six months.
* Patients with unstable angina, ischemic myocardial infarction, or heart failure in the last six months.
* Patients with severe preoperative lung disease (such as pulmonary fibrosis, severe lung abscess, pulmonary heart disease; or with FEV1 less than 50% of the predicted value, PaO2 ≤ 60 mmHg, PaCO2 > 50 mmHg).
* Patients with poorly controlled preoperative hypertension or diabetes mellitus.
* Patients with a past history of dementia, psychosis, or other neurological disorders.
* Patients undergoing concurrent treatment for other surgical conditions.
* Patients taking sedatives, antidepressants, or hormonal medications.
* Patients with chronic pain, alcoholism, or drug dependence.
* Patients who are pregnant or breastfeeding
* Patients with other potentially serious medical conditions.
* Patients who are unable to understand Mandarin or Cantonese.
* Patients who participated in other clinical trials in the past 3 months
* Patients who refuse to participate in the study or sign the informed consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative 48-h analgesic efficacy at cough | Leave the PACU (T0), postoperative 6 hours (T1)、postoperative 12 hours (T2)、 postoperative 24 hours (T3)、 postoperative 36 hours (T4) and postoperative 48 hours (T5).
  The primary outcome is to compare the overall postoperative 48-h analgesic efficacy with cough as indicated by the cumulative area under curve (AUC) for the NRS over the 48-h period using the trapezoidal rule;

SECONDARY OUTCOMES:
Postoperative 48-h analgesic efficacy at rest | Leave the PACU, postoperative 6 hours、postoperative 12 hours、 postoperative 24 hours、 postoperative 36 hours and postoperative 48 hours .
  Compare the overall postoperative 48-h analgesic efficacy at rest as indicated by the cumulative area under curve (AUC) for the NRS over the 48-h period using the trapezoidal rule;
Postoperative quality of recovery | Postoperative 24 hours 、postoperative 48 hours
  Quality of recovery-15 (QoR-15) over the first postoperative 24 and 48 hours.
Postoperative pulmonary complications | From the time of leaving the PACU until the time of the first occurrence of pulmonary complications or the time of death from any cause, whichever came first, assessed up to 30 days.
  Postoperative pulmonary complications are defined as a series of respiratory abnormalities that occur in patients after thoracoscopically assisted lobectomy. These complications may include, but are not limited to: prolonged oxygenation, pulmonary atelectasis, respiratory failure, ARDS, postoperative pneumonia, pleural effusion, pneumothorax, bronchospasm, aspiration pneumonia, and unplanned new or prolonged invasive mechanical ventilation.
The 48-hour postoperative rescue analgesia rate | First 48 hours postoperatively
  The 48-hour postoperative rescue analgesia rate was defined as the percentage of patients requiring additional analgesic medication due to inadequate pain control (NRS score ≥4 at rest) during the 48-hour postoperative period as a proportion of the total number of patients in the group.
Postoperative analgesic failure | First 48 hours postoperatively
  Postoperative analgesic failure was defined as that during postoperative period, the patient uses a pain pump for pain control, and even after implementing rescue analgesic measures, the patient's resting NRS score remains ≥4, or the NRS score during activities (such as coughing) remains ≥7. This indicates that the pain control has not achieved the expected effect and is considered analgesia failure.
Patient satisfaction with postoperative pain ratings | First 48 hours postoperatively
  Patients' satisfaction with analgesic effect will be assessed using Likert scales, where 1 = extremely dissatisfied, 2 = somewhat dissatisfied, 3 = neutral, 4 = somewhat satisfied, and 5 = extremely satisfied
Time to resume | From the time of leaving the PACU until the time to off-bed, bowel movement, and oral intake or the time of death from any cause, whichever came first, assessed up to 7 days.
  The time to off-bed, bowel movement, and oral intake.( measured in days)
The incidence of unplanned ICU admission and reoperation | From the time of leaving the PACU until the time to unplanned ICU admission or reoperation or the time of death from any cause, whichever came first, assessed up to 30 days.
  The incidence of postoperative ICU admissions was defined as the number of patients requiring ICU transfer after surgery as a percentage of the total number of surgical patients over a given period of time.
  The incidence of reoperation was defined as the number of patients requiring additional surgery due to complications or other medical necessities arising after the initial surgery as a percentage of the total number of patients operated on during a given period of time.
The 30d- and 90d- mortality | Of the time from leaving the PACU to the time of postoperative 90day.
  Postoperative 30-day mortality is usually defined as the percentage of patients who die from any cause within 30 days of surgery. This metric is often used to assess the risk of surgery and postoperative recovery.
  Postoperative 90-day mortality, on the other hand, refers to the proportion of patients who die from any cause within 90 days of surgery. This metric is also used to assess surgical outcomes and long-term patient recovery.
Related Adverse Events | First 48 hours postoperatively
  ESPB-related adverse events and opioid-related adverse events ESPB-related adverse events: local infection, local hemorrhage, hematoma, pneumothorax, neurologic injury, local anesthetic toxicity, allergy, epidural anesthesia, total spinal anesthesia, palpitations, perioperative extubation, shock, and death.
  Opioid-related adverse events: postoperative respiratory depression, postoperative nausea and vomiting, postoperative delirium, postoperative constipation and intestinal obstruction, postoperative urinary retention, pruritus, drug abuse, and addiction.

IPD SHARING:
Plan to Share IPD: No